CLINICAL TRIAL: NCT00873743
Title: Postoperative Analgesia and Antihyperalgesia of Tramadol and Acetaminophen Per Oral After Caesarean Section -A Randomised Controlled Trial in Female O-Desmethyl 1 Metabolizers Identified by the Respective Gene-
Brief Title: Analgesia and Antihyperalgesia of Tramadol and Acetaminophen Per Oral After Caesarean Section
Status: Suspended | Type: Observational
Why Stopped: Study was stopped because of ineffectiveness of one investigated Drug
Sponsor: Medical University of Vienna (Other)
Collaborators: University Hospital Schleswig-Holstein (Other)
Responsible Party: Prof. Dr. Stephan Kettner, Department of Anesthesiology, General Inensive Care and Pain Control
Other Study IDs: 31121976-3; Tramal 50mg kapseln 17.688; Zaldiar 37,5mg/325mg
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2009-04-02 (Estimated); Status verified 2009-04

CONDITIONS: Pain; Cesarean Section
Keywords: lower pain intensity with combination drug after cesarian section in first 48h postoperatively
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CYP P450 2D6 metabolizer status
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: 60 women after elective cesarian section
- 2: 60 women after elective cesarian section

SUMMARY:
The aim of this study is to evaluate quality of patient-controlled peroral analgesia after cesarian section using the combination of tramadol and acetaminophen. Research hypothesis is that the combination reduces pain at leg rising more than tramadol alone.

DETAILED DESCRIPTION:
Caesarean section rate is growing in western countries (from 9% by 1980, to 12% by 1990 up to 22-24% in 2002)1.

Pain after Caesarean section involves 2 components, somatic pain from the wound and visceral pain from uterine contractions2. Different mechanisms underlie somatic and visceral pain transmission, at spinal and supraspinal levels, supporting different sensitivity to analgetics2. Pain at rest is usually well controlled by parenteral opioids, while pain induced by movements is less responsive to opioids, requesting higher doses with an increase of side effects3.

Beyond the concern of short term recovery, postoperative pain management has an impact on the risk of developing residual pain after surgery4. Following Caesarean section 18% of patients still suffer from pain 3 months after surgery. 12% still complain after 10 months and for 6% pain is a significant problem, interfering with quality of life and being present daily or almost daily5.

Central sensitization, clinically expressed as hyperalgesia and allodynia, not only contributes to postoperative pain perception, but also is associated with the presence of chronic pain state6.

Aside from tissue damage, the most striking risk factor for developing residual pain seems to be the level of immediate postoperative pain7.

From all published data, it is clear that opioids alone do not completely relieve pain after Caesarean section. Achieving effective acute pain control and minimizing side effects, is best possible by the combination of several analgetics acting through different mechanisms (so called balanced analgesia).8-11

Tramadol is an effective postoperative analgetic, combining mainly µ-opioid and monoaminerg actions with good clinical effect in treating somatic and visceral pain12,13. The postoperative use of tramadol after Caesarean is insufficiently evaluated. Studies evaluate a short period of 614 or 815 hours postoperatively. Metaanalysis sum up a mix of non-gynaecological and gynaecological data together. Edwards et al. 2002 used data from 7 unpublished randomized, double-blind, placebo controlled trials assessing tramadol and acetaminophen with dental, gynaecological and orthopaedic patients15. Moore et al. 199616 used 18 primary trials for data collection, from which only one had been published (Sunshine et al. 1992)14. Thus clear statement of tramadol after Caesarean section is not possible.

NSAID´s, widely used as additives for postoperative pain management, have the inconvenient of gastrointestinal side-effects, increased risk for bleeding and of being secreted in breast milk11. The product prescription of diclofenac, ibuprofen and ketoprufen clearly contraindicates its use by breast feeding women. There is little experience with the use of COXII-Inhibitors by breast feeding women as well. Therefore these drugs are not recommended for postoperative use after Caesarean Section11.

Adding acetaminophen to weak opioids increases the analgetic potency of the opioid component16 and is widely used in obstetrics 14,17. According to the product information acetaminophen is recommended for breast feeding women as no neonatal side-effects have been observed.

Laboratory studies with rats have shown that acetaminophen is able to prevent hyperalgesia and block spinal sensitisation induced by NMDA and Substance P18. The same has been demonstrated in a laboratory setting with tramadol, that is able to prevent and reverse hyperalgesic behaviour in rats19. Furthermore it has been shown that the combination of acetaminophen and tramadol is very effective in inhibiting the quantification of proinflammatory mediators (PGE2, TNFα) in cerebrospinal fluid (CSF) and in preventing the development of hyperalgesia20.

In a human pain model, it could be demonstrated, that combining the drugs enhances antihyperalgesia and leads to supra-additive analgesia21.

In a clinical setting, however, the combination of acetaminophen and tramadol and its effects on postoperative sensitisation and pain has not been evaluated.

Tramadol and acetaminophen are both available for oral administration22. Oral analgetic treatments with various drugs (such as ibuprofen, oxycodone-acetaminophen or metamizol) after Caesarean section have been shown of being superior in terms of patient satisfaction and analgesia compared with parenteral opioid and iv. PCA devices23-25. Parenteral narcotics in general are associated with nausea, vomiting, constipation, pruritus, respiratory depression and sedation. Additionally, PCA devices and their associated stands are cumbersome, which potentially could interfere with newborn infant care. Other drawbacks include the expense and the need for close patient supervision 26-28.

The oral combination of acetaminophen and tramadol in respect of pain control and postoperative sensitization after Caesarean section has not been evaluated yet.

1.2: Study objective: Study objective is to evaluate the analgetic and antihyperalgetic potency of oral tramadol and acetaminophen in combination and alone after Caesarean Section.

In this study the following RESEARCH HYPOTHESIS will be tested:

* Combining tramadol with acetaminophen reduces pain atleg rising more than Tramadol alone
* Combining tramadol with acetaminophen has a dose sparing effect on tramadol
* Side-effects can be reduced by the combination
* The combination reduces the area of Pin-Prick hyperalgesia surrounding the incision more than tramadol alone

ELIGIBILITY:
Inclusion Criteria:

* 18 and 45 years
* ASA-Status 1-2
* BMI 19-29, that are scheduled for planned caesarean section and have given written informed consent

Exclusion Criteria:

* Allergies or hypersensitivities to evaluated drugs
* History of pain syndrome
* Substance abuse
* Preeclampsia or eclampsia
* Deviation from standardised surgical procedure
* Treatment with magnesium sulfate
* Renal or hepatic impairment and deviations from the standardized anaesthetic treatment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female patients postoperatively after cesarian section
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-05 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
VAS-Score at leg rising | 4h, 8h, 24h 48h postoperatively

SECONDARY OUTCOMES:
VAS-Score at rest, nausea, vomitus, sedation, general satisfaction | 4h, 8,h, 24h, 48h postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Kettner, MD, Prof, Principal Investigator — Department of Anesthesiology, General Intensive Care and Pain Control, Medical University Vienna
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria